CLINICAL TRIAL: NCT04009824
Title: Randomized, Double-Blind, Placebo-Controlled, Single-Center, Phase 1 Study in Healthy Volunteers to Evaluate the Safety and Immunogenicity of AGS-v PLUS, a Universal Mosquito-Borne Disease and Mosquito Control Vaccine
Brief Title: Evaluating the Safety and Immunogenicity of AGS-v PLUS, a Universal Mosquito-Borne Disease and Mosquito Control Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: PepTcell Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGS-v PLUS
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Results first posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Mosquito-Borne Infectious Diseases
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: Saline Placebo (Placebo Comparator): Participants received placebo on days 1 and 22 by subcutaneous injection
  Interventions: Biological: Saline Placebo
- Group 2: AGS-v PLUS Non-Adjuvanted (Experimental): Participants received 1012 µg of unadjuvanted AGS-v PLUS vaccine on days 1 and 22 by subcutaneous injection
  Interventions: Biological: AGS-v PLUS Vaccine
- Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo (Experimental): Participants received 1012 µg of AGS-v PLUS and Montanide ISA-51 on day 1 and placebo on day 22 by subcutaneous injection
  Interventions: Biological: AGS-v PLUS Vaccine; Biological: Montanide ISA-51 Adjuvant; Biological: Saline Placebo
- Group 4: AGS-v PLUS + Montanide ISA-51 (Experimental): Participants received 1012 µg of AGS-v PLUS + Montanide ISA-51 on days 1 and 22 by subcutaneous injection
  Interventions: Biological: AGS-v PLUS Vaccine; Biological: Montanide ISA-51 Adjuvant
- Group 5: AGS-v PLUS + Alhydrogel® Adjuvant (Experimental): Participants received 1012 µg of AGS-v PLUS and Alhydrogel® on days 1 and 22 by subcutaneous injection
  Interventions: Biological: AGS-v PLUS Vaccine; Biological: Alhydrogel® Adjuvant

INTERVENTIONS:
Biological: AGS-v PLUS Vaccine — Administered by subcutaneous injection
  Arms: Group 2: AGS-v PLUS Non-Adjuvanted; Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo; Group 4: AGS-v PLUS + Montanide ISA-51; Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Biological: Montanide ISA-51 Adjuvant — Administered by subcutaneous injection
  Arms: Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo; Group 4: AGS-v PLUS + Montanide ISA-51
Biological: Alhydrogel® Adjuvant — Administered by subcutaneous injection
  Arms: Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Biological: Saline Placebo — Administered by subcutaneous injection
  Arms: Group 1: Saline Placebo; Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of AGS-v PLUS, a universal mosquito-borne disease and mosquito control vaccine, in healthy volunteers.

DETAILED DESCRIPTION:
This study will evaluate the safety and immunogenicity of AGS-v PLUS, a universal mosquito-borne disease and mosquito control vaccine, in healthy volunteers.

Participants will be randomly assigned to five groups.

Participants in Group 1 will receive placebo on Days 1 and 22.

Participants in Group 2 will receive unadjuvanted AGS-v PLUS vaccine on Days 1 and 22.

Participants in Group 3 will receive Montanide ISA-51 adjuvanted AGS-v PLUS vaccine on Day 1 and placebo on Day 22.

Participants in Group 4 will receive Montanide ISA-51 adjuvanted AGS-v PLUS vaccine on Days 1 and 22.

Participants in Group 5 will receive Alhydrogel® adjuvanted AGS-v PLUS vaccine on Days 1 and 22.

Participants will be in the study for approximately 12 months. During this time, they will attend several study visits, which may include physical examinations, blood collection, skin biopsies, and a mosquito feeding procedure. Study staff will also follow up with participants by phone several times throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and men who are greater than or equal to 18 and less than or equal to 50 years of age.
* Willingness to complete all study visits and comply with all study requirements.
* A male participant is eligible for the study if he agrees to practicing abstinence or using a condom with spermicide plus an acceptable form of contraception (see inclusion criteria below) being used by any female partner from 4 weeks before study start to 12 weeks after the second vaccine administration.
* A female participant is eligible for this study if she is not pregnant or breast feeding and 1 of the following:

  * Of non-child bearing potential (i.e., women who have had a hysterectomy or tubal ligation, or are postmenopausal, as defined by no menses in greater than or equal to 1 year).
  * Of childbearing potential but agrees to practice effective contraception or abstinence for 4 weeks before study initiation and 12 weeks after the second vaccine administration. Acceptable methods of contraception include a female partner who is the sole sexual partner of the female participant, a male partner who is sterile and is the sole sexual partner of the female participant, or a male partner who uses a condom with spermicide plus 1 or more of the following: 1) implants of levonorgestrel; 2) injectable progestogen; 3) an intrauterine device with a documented failure rate of less than 1%; 4) oral contraceptives; and 5) double barrier method including diaphragm.
* Willing to have samples stored for future research.
* Agrees to abstain from alcohol intake for 24 hours before each study visit.
* Agrees to not donate blood or blood products throughout the study.
* Score greater than or equal to 70% on comprehension quiz at screening

Exclusion Criteria:

* Participant has any underlying or current medical condition, which, in the opinion of the Investigator, would interfere with the participation in the study.
* Individual with body mass index (BMI) less than or equal to 18 and greater than or equal to 40.
* Participants who have a clinically significant (as determined by the PI or designee) baseline Grade 1 or greater toxicity, or any Grade 2 or greater toxicity (regardless of clinical significance) by the toxicity table.
* Receipt of blood or blood products including immunoglobulin within 3 months before enrollment.
* Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) before enrollment.
* Receipt of any unlicensed vaccine within 6 months before enrollment.
* Participated in study NCT03055000 testing safety and immunogenicity of AGS-v.
* Self-reported or known history of alcoholism or drug abuse within 6 months before enrollment.
* Self-reported or known history of psychiatric or psychological issues that require treatment and are deemed by the PI or designee to be a contraindication to protocol participation.
* History of a previous severe allergic reaction with generalized urticaria, angioedema, anaphylaxis or anaphylactoid reaction.
* Any condition or event that, in the judgment of the PI or designee, is a contraindication to protocol participation or impairs the volunteer's ability to give informed consent.
* Known allergy to any vaccine component, including adjuvants.
* History of severe immunization reaction.
* Severe allergic reaction to mosquito bites (anaphylaxis)
* Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days before study vaccination
* Have taken high-dose inhaled corticosteroids* within 30 days before each study vaccination (* High-dose defined per age as using inhaled high dose per reference chart: https://www.nhlbi.nih.gov/sites/default/files/media/docs/asthma_qrg_0_0.pdf)
* Received or plan to receive a licensed, live vaccine within 30 days before or after the study vaccination
* Received or plan to receive a licensed, inactivated vaccine within 14 days before or after study vaccination
* Serologic evidence of infection with HIV, hepatitis B virus, or hepatitis C virus
* Ongoing chronic skin condition, or acute skin condition at the time of vaccination or mosquito feeding, except for mild eczema.
* History of keloid formation after previous biopsies, lacerations, abrasions, surgeries, or other skin procedures (e.g., cosmetic piercings) that are deemed by the PI or designee to be a contraindication to protocol participation.
* Pregnancy, breastfeeding, or planning to become pregnant up to one month after mosquito feeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B. Laurens, MD, MPH, Principal Investigator — University of Maryland, Baltimore; Matthew J. Memoli, MD, MS, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Started | 10 | 10 | 11 | 10 | 10
Completed | 8 | 7 | 6 | 8 | 7
Not Completed | 2 | 3 | 5 | 2 | 3
Not completed — COVID-19 pandemic restriction/closure | 2 | 3 | 5 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant | Total
Number analyzed (Participants) | 10 | 10 | 11 | 10 | 10 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 11 | 10 | 10 | 51
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 6 | 5 | 5 | 21
  Male | 8 | 7 | 5 | 5 | 5 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 10 | 10 | 10 | 10 | 9 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 5 | 4 | 1 | 21
  White | 3 | 4 | 4 | 5 | 7 | 23
  More than one race | 0 | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 11 | 10 | 10 | 51

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Severity of Treatment Emergent Adverse Events (AEs) by Grade
Description: A treatment emergent adverse event is any untoward medical occurrence in a human subject that manifest after administration of the study treatment, whether or not considered related to the treatment. AE severity was graded using FDA Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, September 2007 or the following grading scale:
  Grade 1 (Mild) Events causing no or minimal interference with daily activity and not requiring medical intervention Grade 2 (Moderate) Events causing greater than minimal interference with daily activity but not requiring medical intervention Grade 3 (Severe) Events causing inability to perform daily activity and/or requiring medical intervention Grade 4 (Potentially Life-Threatening)* Events causing inability to perform basic self-care functions OR medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death Grade 5 (Death) Events causing death
Time Frame: 1 year
Population: All participants who started the study
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 10 | 10 | 11 | 10 | 10
Participants
  Grade 1 | 7 | 8 | 10 | 8 | 4
  Grade 2 | 3 | 2 | 4 | 7 | 1
  Grade 3 | 0 | 0 | 4 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Mean log10 Titer in Serum AGS-v PLUS Specific Immunoglobulin Titers
Description: Mean log10 titer in serum AGS-v PLUS specific immunoglobulin E (IgE), immunoglobulin G (IgG), and immunoglobulin M (IgM) titers were assessed using enzyme-linked immunosorbent assay (ELISA)
Time Frame: Day 43
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: log10 titer
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 8 | 7
log10 titer
  IgE | 2.5399 (0.1666) | 2.4628 (0.1606) | 2.4915 (0.1552) | 2.4414 (0.1606) | 2.5058 (0.1466)
  IgG | 3.3425 (0.7442) | 3.8098 (0.4761) | 3.7625 (0.6941) | 4.1428 (0.4795) | 3.3863 (0.3979)
  IgM | 3.0480 (0.3253) | 3.0465 (0.3513) | 3.3010 (0.4430) | 3.4840 (0.5158) | 3.1993 (0.4856)

3. Primary Outcome: Mean log10 Fold Change in Serum AGS-v PLUS Specific Immunoglobulin Titer
Description: Mean log10 fold change in serum AGS-v PLUS specific immunoglobulin G (IgG), immunoglobulin M (IgM) and immunoglobulin E (IgE) titers from day 1 to day 43 assessed using enzyme-linked immunosorbent assay (ELISA). The fold change from day 1 to day 43 is calculated by dividing the antibody titer for a specific isotype i.e. IgE at day 43 by the titer at day 1. In order to stabilize the variance, the log10 of the fold change was used in the analyses.
Time Frame: Day 1 and Day 43
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: log10 fold change
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 8 | 7
log10 fold change
  IgE | 0.0553 (0.1563) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000)
  IgG | -0.0151 (0.0553) | 0.2432 (0.2250) | 1.1274 (0.7249) | 1.3033 (0.7104) | 0.5336 (0.5084)
  IgM | -0.0121 (0.0963) | 0.1826 (0.2759) | 0.2988 (0.4061) | 0.5530 (0.4568) | -0.0114 (0.2509)

4. Primary Outcome: Mean log10 Concentration in Th1 and Th2 Cytokine Responses
Description: Mean log10 concentration in Th1 (IFN-gamma) and Th2 (IL-4) cytokine responses after in vitro exposure of peripheral blood mononuclear cells (PBMCs) with AGS-v PLUS antigens assessed using enzyme-linked immunosorbent assay (ELISA)
Time Frame: Day 43
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 8 | 7
pg/ml
  IFN-gamma | 0.1909 (0.6279) | 1.4052 (1.1236) | 1.6730 (0.9671) | 1.5934 (0.8151) | 1.5007 (1.1989)
  IL4 | -2.1753 (1.2352) | -2.3499 (1.2972) | -0.8076 (2.2295) | -0.7952 (1.7543) | 0.4814 (1.5686)

5. Primary Outcome: Mean log10 Fold Change in Th1 and Th2 Cytokine Responses
Description: Mean log10 fold change in Th1 (IFN-gamma) and Th2 (IL-4) cytokine responses after in vitro exposure of peripheral blood mononuclear cells (PBMCs) with AGS-v PLUS antigens from day 1 to day 43 assessed using enzyme-linked immunosorbent assay (ELISA). The fold change from day 1 to day 43 is calculated by dividing the antigen titer for a specific isotype i.e. IFN-gamma at day 43 by the titer at day 1. In order to stabilize the variance, the log10 of the fold change was used in the analyses.
Time Frame: Day 1 and Day 43
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: log10 fold change
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 7 | 7 | 6 | 8 | 7
log10 fold change
  IFN-gamma | -1.0560 (1.2765) | 0.7983 (1.6906) | 1.1645 (1.7015) | 1.0486 (1.1661) | 0.9757 (1.4482)
  IL4 | 0.3529 (0.9338) | 0.0576 (0.1523) | 1.6160 (1.9909) | 1.4378 (1.4169) | 3.2786 (1.5472)

6. Secondary Outcome: Mean log10 Titer in Serum AGS-v PLUS Specific Immunoglobulin Titer
Description: Mean log10 titer in serum AGS-v PLUS specific immunoglobulin G (IgG), immunoglobulin M (IgM) and immunoglobulin E (IgE) titers seven days after mosquito feeding assessed using enzyme-linked immunosorbent assay (ELISA)
Time Frame: Day 50
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: log10 titer
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 6
log10 titer
  IgE | 2.502 (0.1362) | 2.4628 (0.1606) | 2.4915 (0.1552) | 2.4074 (0.1475) | 2.4915 (0.1552)
  IgG | 3.3322 (0.7409) | 3.7976 (0.4694) | 3.8225 (0.7273) | 4.4132 (0.4667) | 3.4214 (0.3945)
  IgM | 3.0461 (0.3381) | 3.0263 (0.3157) | 3.3270 (0.4327) | 3.7576 (0.2931) | 3.2060 (0.4878)

7. Secondary Outcome: Mean log10 Fold Change in Serum AGS-v PLUS Specific Immunoglobulin Titer
Description: Mean log10 fold change in serum AGS-v PLUS specific immunoglobulin G (IgG), immunoglobulin M (IgM) and immunoglobulin E (IgE) titers from day 1 to day 50 assessed using enzyme-linked immunosorbent assay (ELISA). The fold change from day 1 to day 50 is calculated by dividing the antibody titer for a specific isotype i.e. IgE at day 50 by the titer at day 1. In order to stabilize the variance, the log10 of the fold change was used in the analyses.
Time Frame: Day 1 and Day 50
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: log10 fold change
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 6
log10 fold change
  IgE | 0.0174 (0.0491) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0161 (0.0395) | 0.0000 (0.0000)
  IgG | -0.0254 (0.0552) | 0.2309 (0.2134) | 1.1874 (0.7482) | 1.4047 (0.8537) | 0.5295 (0.4994)
  IgM | -0.0139 (0.0967) | 0.1623 (0.2306) | 0.3247 (0.3746) | 0.6928 (0.5505) | 0.0204 (0.3250)

8. Secondary Outcome: Mean log10 Fold Change in Serum AGS-v PLUS Specific Immunoglobulin Titer
Description: Mean log10 fold change in serum AGS-v PLUS specific immunoglobulin G (IgG), immunoglobulin M (IgM) and immunoglobulin E (IgE) titers seven days after mosquito feeding assessed using enzyme-linked immunosorbent assay (ELISA). The fold change from day 43 to day 50 is calculated by dividing the antibody titer for a specific isotype i.e. IgE at day 50 by the titer at day 43. In order to stabilize the variance, the log10 of the fold change was used in the analyses.
Time Frame: Day 43 and Day 50
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: log10 fold change
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 6
log10 fold change
  IgE | -0.0379 (0.1072) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0161 (0.0395) | 0.0000 (0.0000)
  IgG | -0.0103 (0.0102) | -0.0122 (0.0328) | 0.0601 (0.0705) | 0.1256 (0.0968) | 0.0701 (0.0705)
  IgM | -0.0018 (0.0459) | -0.0202 (0.0674) | 0.0260 (0.1005) | 0.0200 (0.1188) | 0.0273 (0.1175)

9. Secondary Outcome: Mean log10 Concentration in Th1 and Th2 Cytokine Responses
Description: Mean log10 concentration in Th1 (IFN-gamma) and Th2 (IL-4) cytokine responses after in vitro exposure of peripheral blood mononuclear cells (PBMCs) with AGS-v PLUS antigens seven days after mosquito feeding assessed using enzyme-linked immunosorbent assay (ELISA)
Time Frame: Day 50
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 6
pg/ml
  IFN-gamma | 0.3648 (0.9467) | 0.7095 (1.1809) | 1.9669 (0.3134) | 1.7539 (0.6509) | 1.8744 (1.0427)
  IL4 | -2.2435 (1.1230) | -2.3313 (1.3465) | -0.8640 (2.1660) | -0.7668 (1.6473) | -0.7570 (2.2994)

10. Secondary Outcome: Mean log10 Fold Change in Th1 and Th2 Cytokine Responses
Description: Mean log10 fold change in Th1 (IFN-gamma) and Th2 (IL-4) cytokine responses after in vitro exposure of peripheral blood mononuclear cells (PBMCs) with AGS-v PLUS antigens from day 1 to day 50 assessed using enzyme-linked immunosorbent assay (ELISA). The fold change from day 1 to day 50 is calculated by dividing the antigen titer for a specific isotype i.e. IFN-gamma at day 50 by the titer at day 1. In order to stabilize the variance, the log10 of the fold change was used in the analyses.
Time Frame: Day 1 and Day 50
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: log10 fold change
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 7 | 7 | 6 | 6 | 6
log10 fold change
  IFN-gamma | -0.8572 (1.2638) | 0.1025 (1.2759) | 1.4584 (0.9659) | 1.2067 (1.3654) | 1.5043 (1.0085)
  IL4 | 0.6819 (1.1847) | 0.0762 (0.2016) | 1.5597 (1.9207) | 1.2638 (1.3559) | 2.0330 (2.2454)

11. Secondary Outcome: Mean log10 Fold Change in Th1 and Th2 Cytokine Responses
Description: Mean log10 fold change in Th1 (IFN-gamma) and Th2 (IL-4) cytokine responses after in vitro exposure of peripheral blood mononuclear cells (PBMCs) with AGS-v PLUS antigens seven days after mosquito feeding assessed using enzyme-linked immunosorbent assay (ELISA). The fold change from day 43 to day 50 is calculated by dividing the antigen titer for a specific isotype i.e. IFN-gamma at day 50 by the titer at day 43. In order to stabilize the variance, the log10 of the fold change was used in the analyses.
Time Frame: Day 43 and Day 50
Population: All participants who completed the study and had sample available
Measure: Mean (Standard Deviation); unit: log10 fold change
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 6
log10 fold change
  IFN-gamma | 0.1739 (1.0779) | -0.6957 (1.0983) | 0.2939 (0.8593) | 0.2227 (1.0546) | 0.0855 (0.1705)
  IL4 | -0.0682 (1.3204) | 0.0186 (0.0493) | -0.0563 (0.1880) | -0.6533 (1.2554) | -1.1923 (1.8252)

12. Secondary Outcome: Mean Days of Mosquitoes Survival Post Feeding
Description: Mean days of Aedes aegypti and Aedes albopictus female mosquitoes survival post feeding on study participants
Time Frame: Day 43
Population: All participants who completed the study and underwent mosquito feeding
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 6
Days
  Aedes aegypti | 6.912 (0.247) | 6.757 (0.522) | 6.783 (0.299) | 6.733 (0.301) | 6.850 (0.251)
  Aedes albopictus | 6.775 (0.282) | 6.671 (0.446) | 6.750 (0.446) | 6.817 (0.360) | 6.500 (0.514)

13. Secondary Outcome: Mean Number of Eggs Laid Per Mosquito Post Feeding
Description: Mean number of eggs laid per Aedes aegypti and Aedes albopictus female mosquito post feeding on study participants
Time Frame: Day 43
Population: All participants who completed the study and underwent mosquito feeding
Measure: Mean (Standard Deviation); unit: eggs per mosquito
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 6
eggs per mosquito
  Aedes aegypti | 41.937 (23.112) | 48.019 (13.618) | 58.865 (19.524) | 50.306 (24.500) | 44.314 (17.278)
  Aedes albopictus | 13.140 (8.355) | 7.225 (7.687) | 6.566 (7.151) | 5.114 (7.394) | 7.866 (8.581)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Tracked during clinic visits and follow up phone calls
Arm/Group | Group 1: Saline Placebo | Group 2: AGS-v PLUS Non-Adjuvanted | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo | Group 4: AGS-v PLUS + Montanide ISA-51 | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 8/10 | 11/11 | 9/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Saline Placebo (N=10) | Group 2: AGS-v PLUS Non-Adjuvanted (N=10) | Group 3: AGS-v PLUS + Adjuvant Montanide ISA-51 + Placebo (N=11) | Group 4: AGS-v PLUS + Montanide ISA-51 (N=10) | Group 5: AGS-v PLUS + Alhydrogel® Adjuvant (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 5 (9) | 1 (2) | 4 (7) | 4 (9) | 1 (1)
Application site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site swelling (General disorders) | 2 (2) | 1 (2) | 2 (3) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (3) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Endocrine disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polycystic ovaries (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria papular (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site bruising (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site induration (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vaccination site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaccination site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04009824/Prot_SAP_000.pdf